CLINICAL TRIAL: NCT04427124
Title: Impact of Multidisciplinary Critical Limb Ischemia Team on the Utilization of Vascular Studies, Patient Management, AMPutation and Long-term Outcomes: The CLI-AMP Registry
Brief Title: The CLI-AMP Registry
Acronym: CLI-AMP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hendrick Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Joji Varghese, Principal Investigator, Hendrick Medical Center
Other Study IDs: CA10142019
Record Dates: First submitted 2020-05-06; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Critical Limb Ischemia; Peripheral Arterial Disease; Amputation
Keywords: Critical Limb Ischemia; Peripheral Arterial Disease; Amputation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: Patients admitted into the hospital will receive care based on a multidisciplinary team approach and Institutional critical limb ischemia protocol.
  Interventions: Other: Multidisciplinary Team Based Care Model
- Retrospective: A retrospective analysis of all patients with CLI admitted to the hospital from 2017-2019 will serve as a baseline comparator for overall CLI care and long-term mortality out to 2 years will be analyzed in the retrospective cohort using the national death index. Patients will be identified by the following ICD codes: 440.22 (ASVD of extremities with rest pain), 440.23 (ulceration), and 440.24 (gangrene).

INTERVENTIONS:
Other: Multidisciplinary Team Based Care Model — All prospective patients admitted into the study will receive care based on multidisciplinary team collaboration and an institutional protocol for critical limb ischemia.
  Groups: Prospective

SUMMARY:
Single-center, observational registry study with a prospective and retrospective arm to evaluate the impact of multidisciplinary CLI teams and protocol on amputation rates, vascular studies, revascularization, in-hospital and long-term outcomes.

DETAILED DESCRIPTION:
It is well known from large Medicare and National Inpatient Sample databases that vascular evaluations in patients with critical limb ischemia (CLI) and at risk for amputations remains extremely low. However, this data is largely pulled from the early 2000s with a scarcity in studies from this recent decade. A recent study showed that Medicare patients from 2011 showed that 23% of patients received primary major amputation. In a recent retrospective analysis preformed at this institution, all amputation patients from 2011-2017 were evaluated for vascular work up and long-term mortality. This cohort included 698 patients with 1009 amputated specimens (major and minor). This means that this institution is preforming around 140 amputations per year, which can be considered unacceptably high. Only 50% received any form of vascular study (ankle-brachial index, doppler ultrasound, and computed tomography angiography) within the year prior to amputation. Furthermore, only 30% of patients received an angiogram within the year prior to amputation. In addition, all major amputations received histopathological analysis, which confirmed that 62% the specimens were graded with severe atherosclerosis. Even in this present decade, with the knowledge that CLI patients are not receiving proper evaluation and treatment leading to amputation which is associated with extreme mortality rates and a large economic burden, health care facilities are not improving their care.

Multidisciplinary teams are a recommendation from the American Heart Association/American College of Cardiology guidelines for managing peripheral vascular disease. Multidisciplinary team approaches in other cardiovascular diseases, such as structural heart disease, has long been validated. Literature regarding the implementation of "CLI Teams" remains scarce and not widely adopted. However, institutions that have implemented a CLI Team that engages with specialists from multiple disciplines have shown successful decrease in amputation rates and increases in vascular evaluations and revascularization in these patients. The goal for this study is to establish a hospital-based, physician and nurse led, multidisciplinary team to deliver comprehensive care to CLI patients. We believe it is important to document the experience of building a CLI Team and care protocols to provide insight and validated data for other programs to implement. The multidisciplinary team will include vascular interventionalists, hospitalists, podiatry, wound care, infectious disease, nephrology, orthopedics, pharmacists, emergency department physicians, mid-level providers, nursing staff, and vascular technologists. The ultimate goal is amputation prevention and wound healing through comprehensive vascular care and data driven patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* CLI of the lower extremity
* Willingness and ability to participate in the study and meet follow-up requirements

Exclusion Criteria:

* Pregnancy
* <18 years of age
* Incarcerated patients
* Patients who receive amputations due to trauma or cancer
* Wound, gangrene, or amputation of the upper extremities
* Unwillingness or inability to participate in the study and meet follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Critical Limb Ischemia
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the number of major amputations within the hospital | 2 years
  Decreased percentage
Change in in-hospital and long-term mortality rates | 2 years

SECONDARY OUTCOMES:
Change in the percentage of non-invasive vascular evaluations in patients with CLI and at risk for amputation (ABI, DUS, CTA) | 2 years
Change in percentage of patients receiving invasive angiogram and revascularization (Endovascular or Surgical). | 2 years
Change in wound healing | 2 years
  Decrease in Rutherford Classification
Change in hospital length of stay | 2 years
  Decrease in days

IPD SHARING:
Plan to Share IPD: No